CLINICAL TRIAL: NCT02624232
Title: Long-term Outcome in Patients Operated for Congenital Anorectal Malformations
Brief Title: Long-term Outcome in Patients With Anorectal Malformations
Acronym: LOPAM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thomas Bjørsum-Meyer, M.D.,ph.d-student, Odense University Hospital
Other Study IDs: S-20140017
Record Dates: First submitted 2015-11-17; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Anorectal Malformation
Keywords: Anorectal malformation; Anorectal atresia; anorectal stenosis; Follow-Up Studies
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with anorectal malformations: Participants are identified through relevant diagnostic codes in ICD-10(Q 42) and ICD-9(75.120, 75.121) in patients which underwent surgery for ARM in the years 1985-2005 are included if informed consent is obtained.
  Relevant questionnaires regarding symptoms and QoL are completed before the following examinations:anorectal manometry, endoanal ultrasonography, pudendal nerve conduction velocity, colon transit time, Magnetic resonans(MR)-scan of the pelvis and uroflowmetry.

SUMMARY:
Background Anorectal malformations(ARM) are rare and cover congenital defective development of rectum.

ARM include a range of congenital conditions and may in varying degrees involve the anorectum. A significant part have malformations in other organs mainly the urinary tract.

In the vast majority ARM are recognized at birth by lack of a normal anus. The primary approach is construction of a stoma and subsequent reconstruction. Bowel continuity is typical restored after 4-6 months.

Many patients experience abnormal bowel function later on and affected quality of life(QoL).

Aim

The primary objective is to assess the patient-related outcome 10-30 years after surgery for ARM and to see if it related to existing damage to anorectum and bowel function. The secondary objective is to identify problems with bowel function which may be treated medically or by surgery to improve bowel function and QoL. To obtain the necessary knowledge the study is divided in the following sub-projects:

1. Assessment of bowel function and QoL through relevant questionnaires
2. Examine sphincter anatomy and function through rectal ultrasound, magnetic resonans(MR)-scan of the pelvis and anal manometry. Bowel function is assessed through colonic transit time. Screening for urinary tract problems with uroflowmetry.

Methods Participants are identified through relevant diagnostic codes(Q 42) and patients which underwent surgery for ARM in the years 1985-2005 are included if informed consent is obtained.

Relevant questionnaires regarding symptoms and QoL are completed before the following examinations:

* Anal manometry
* Anal ultrasound
* Pudenda conduction velocity
* Colonic transit time
* Magnetic resonans(MR)-scan of lower abdomen and pelvis
* Uroflowmetry

Bowel function and QoL is assessed in both children and adults with relevant validated questionnaires.

Perspective No danish studies and only a few foreign investigate the relationship between anatomy/physiology and quality of life after surgery for anorectal malformations.

The investigators believe the study and included comprehensive examinations will clarify the causes of functional problems after surgery for anorectal malformations. Results of questionnaires regarding symptoms, disease-specific-and general quality of life offer a unique opportunity for targeted treatment to improve symptoms and QoL in patients with ARM.

DETAILED DESCRIPTION:
Aim

Endpoints The primary endpoints are outcome 10-30 years after surgery for anorectal malformations and to see if it is related to existing altered anatomy, anorectal function and intestinal passage.

The secondary endpoints is to identify bowel function problems which can be treated by medicine or surgery to improve patients bowel function and quality of life.

To obtain the necessary knowledge the study will be divided in the following

Sub-projects:

1. Evaluation of bowel function and quality of life with relevant questionnaire.
2. Examine anorectal anatomy and function with anal ultrasound, Magnetic resonans(MR)-scan of the small pelvis and anal manometry. Overall bowel function is examined with colonic transit time. Screening for urinary problems with urodynamic testing.

Background Anorectal malformations(ARM) cover a wide spectrum of congenital disorders seen in both sexes and may also involve the urinary tract and genitals. It occurs in 1/2500 of newborns with a slight predominance in boys and 2/3 have accompanying anomalies. ARM form as an abnormal development of the hindgut which later forms the descending colon, rectum, anus, bladder and urethra. This explains frequent recurrence of accompanying malformations in the urinary tract.

The reason for the development of ARM is unknown. The etiology is probably multifactorial including both heredity and environment. A chromosomal anomaly is found among 5% of patients with ARM and Trisomy 21 being most common. Possible risk factors is maternal fever in the first trimester, industrial exposure to solvents, paternal smoking, maternal obesity and diabetes.

Accompanying anomalies often involve more organ systems. The mortality among patients with ARM is 10-20 % and is primary seen with high malformations having most severe associated anomalies including cardiac.

Previously the classification of ARM was based upon sex and the position of rectum relative to the levator ani muscle in high, intermediate and low(Wingspread classification). Pena and colleagues suggested in the mid 90s a classification system based on the presence of a fistula. Later the Krickenbeck classification system was introduced which classify ARM based on appearance, surgical approach and symptoms.

The classic surgical approach consists of an early divergent stoma, later a surgical correction and finally closure of the stoma.The classic surgical treatment of intermediate and high ARM was an abdominoperineal pull-through technique. Later Pena and colleagues introduced posterior sagittal anorectal plasty(PSARP). PSARP was adapted at Odense University hospital in 1994 and still the preferred surgical approach. Last laparoscopic assisted anorectal pull-through(LAARP) has been introduced but has not gain common accept.

Functional problems after ARM is primary fecal incontinence for high and constipation for low malformations.Treatment is primary medical or dietetic regulation of the bowel and in treatment-resistent cases anal irrigation and appendicostomy and antegrade colonic irrigation. Sometimes a permanent stoma may be needed.

Different imaging techniques and physiological measures have been used to clarify the anatomy and bowel function after surgical correction of ARM.

MRI(magnetic resonance imaging) of the pelvis has shown differences in patients with constipation and fecal incontinence after surgery for ARM. MRI provides useful information regarding pelvic musculature, colonic anatomy and other accompanying disorders. Anal ultrasound and manometry are useful to evaluate the anatomy and function of the anal sphincter. Scar tissue formation and defects in the anal sphincter are correlated to pressure in the anal canal and fecal incontinence.

A recent technique to evaluate the anorectal neuromuscular function is High Resolution Anorectal Manometry(HRAM). HRAM has previously proven to be more accurate in displaying anorectal anatomy compared to water-perfused manometry. Colonic transit time provides information about motility disorders and in patient with constipation colonic hypomobility is observed.

Pudendal nerve conduction velocity can be useful in evaluating fecal incontinence and delayed conduction velocity observed.

An essential issue regarding ARM is quality of life(QoL). A literature review by Witvliet and colleagues showed that only 20% of published studies used validated questionnaires.(30) Nine of 30 included studies on QoL were performed on an adult population. Poyet and colleagues found Health Related Quality of Life(HRQoL) was affected among patient aged one to four years compared to a control group after surgery for ARM. Hartmann et al. found no changes during a period of three years in an adult population. Women, older patients, patients with other defects and patients with a stoma reported reduced QoL.

Statistics It is mainly a descriptive study and therefore power calculation is neither possible nor relevant. In recruitment period an average of 10 patients have undergone surgery annually at the University Hospital of Odense. The investigators expect more than 50% of patients will participate and the population would be one of the largest yet seen. It will be possible to prove clinical relevant differences(20%) or correlations between different operative techniques. Further more it is possible to prove correlations between symptoms and outcome of different imaging techniques, examinations and questionnaires.

Questionnaires Symptoms and QoL are assessed with questionnaires. Bowel function after surgery for anorectal malformations is evaluated with the Krickenbeck Classification. In adults also with Wexner's Incontinence score and Cleveland Clinic Constipation Score(CCCS).

Disease-specific QoL in adults is assessed with Fecal Incontinence QoL(FIQL) and general QoL with the EQ-5D-5L. In participants below 18 years of age general QoL is assessed with Strenght and Difficulties Questionnaire(SDQ).

Urinary function and impact on quality of life in adults is evaluated with International Consultation on Incontinence Modular Questionnaire - Female Lower Urinary Tract Symptoms(ICIQ-FLUTS) and International Consultation on Incontinence Modular Questionnaire - Male Lower Urinary Tract Symptoms(ICIQ-MLUTS).

Sexual function is assessed with International Index of Erectile Dysfunction(IIEF) and in women with Female Sexual Function Index(FSFI).

Only Danish version of questionnaires are used.

Course plan The project will run for three years(2014-2017) and it is intended that all subjects have completed examinations before July 2016. The participants will be asked to fill in the different questionnaire regarding bowel habits, symptoms and QoL. There are planned hospitalization for participants for two days and they may stay overnight at the patient hotel or at home. Initially medical history is obtained, clinical examination performed and questionnaires collected.

Perspective No danish studies and only a few foreign investigate the relationship between anatomy/physiology and quality of life after surgery for anorectal malformations.

The investigators believe the study and included comprehensive examinations will clarify the causes of functional problems after surgery for anorectal malformations. Results of questionnaires regarding symptoms, disease-specific-and general quality of life offer a unique opportunity for targeted treatment to improve symptoms and QoL in patients with ARM.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for anorectal malformations

Exclusion Criteria:

* Severe mental disability

Ages: 10 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants are born with anorectal malformations and subjected to surgery at the Odense University Hospital during the period 1985 - 2004.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between anorectal pathoanatomy and gastrointestinal symptoms/quality of life | Up to 6 years

SECONDARY OUTCOMES:
Correlation between gastrointestinal symptoms and quality of life | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Study Director — Research unit for Surgery

REFERENCES:
- [Background] Levitt MA, Pena A. Anorectal malformations. Orphanet J Rare Dis. 2007 Jul 26;2:33. doi: 10.1186/1750-1172-2-33. PMID 17651510
- [Background] Cuschieri A; EUROCAT Working Group. Descriptive epidemiology of isolated anal anomalies: a survey of 4.6 million births in Europe. Am J Med Genet. 2001 Oct 15;103(3):207-15. doi: 10.1002/ajmg.1532.abs. PMID 11745992
- [Background] Mittal A, Airon RK, Magu S, Rattan KN, Ratan SK. Associated anomalies with anorectal malformation (ARM). Indian J Pediatr. 2004 Jun;71(6):509-14. doi: 10.1007/BF02724292. PMID 15226560
- [Background] Lowry RB, Sibbald B, Bedard T. Stability of prevalence rates of anorectal malformations in the Alberta Congenital Anomalies Surveillance System 1990-2004. J Pediatr Surg. 2007 Aug;42(8):1417-21. doi: 10.1016/j.jpedsurg.2007.03.045. PMID 17706507
- [Background] Jenetzky E. Prevalence estimation of anorectal malformations using German diagnosis related groups system. Pediatr Surg Int. 2007 Dec;23(12):1161-5. doi: 10.1007/s00383-007-2023-6. PMID 17929037
- [Background] Herman RS, Teitelbaum DH. Anorectal malformations. Clin Perinatol. 2012 Jun;39(2):403-22. doi: 10.1016/j.clp.2012.04.001. PMID 22682388
- [Background] Marcelis C, de Blaauw I, Brunner H. Chromosomal anomalies in the etiology of anorectal malformations: a review. Am J Med Genet A. 2011 Nov;155A(11):2692-704. doi: 10.1002/ajmg.a.34253. Epub 2011 Oct 11. PMID 21990113
- [Background] Wijers CH, de Blaauw I, Marcelis CL, Wijnen RM, Brunner H, Midrio P, Gamba P, Clementi M, Jenetzky E, Zwink N, Reutter H, Bartels E, Grasshoff-Derr S, Holland-Cunz S, Hosie S, Marzheuser S, Schmiedeke E, Cretolle C, Sarnacki S, Levitt MA, Knoers NV, Roeleveld N, van Rooij IA. Research perspectives in the etiology of congenital anorectal malformations using data of the International Consortium on Anorectal Malformations: evidence for risk factors across different populations. Pediatr Surg Int. 2010 Nov;26(11):1093-9. doi: 10.1007/s00383-010-2688-0. PMID 20730541
- [Background] Zwink N, Jenetzky E, Brenner H. Parental risk factors and anorectal malformations: systematic review and meta-analysis. Orphanet J Rare Dis. 2011 May 17;6:25. doi: 10.1186/1750-1172-6-25. PMID 21586115
- [Background] Cuschieri A; EUROCAT Working Group. Anorectal anomalies associated with or as part of other anomalies. Am J Med Genet. 2002 Jun 15;110(2):122-30. doi: 10.1002/ajmg.10371. PMID 12116249
- [Background] Rintala RJ, Pakarinen MP. Imperforate anus: long- and short-term outcome. Semin Pediatr Surg. 2008 May;17(2):79-89. doi: 10.1053/j.sempedsurg.2008.02.003. PMID 18395657
- [Background] Stephens FD. Wingspread anomalies, rarities, and super rarities of the anorectum and cloaca. Birth Defects Orig Artic Ser. 1988;24(4):581-5. No abstract available. PMID 3228583
- [Background] Pena A, Hong A. Advances in the management of anorectal malformations. Am J Surg. 2000 Nov;180(5):370-6. doi: 10.1016/s0002-9610(00)00491-8. PMID 11137690
- [Background] Holschneider A, Hutson J, Pena A, Beket E, Chatterjee S, Coran A, Davies M, Georgeson K, Grosfeld J, Gupta D, Iwai N, Kluth D, Martucciello G, Moore S, Rintala R, Smith ED, Sripathi DV, Stephens D, Sen S, Ure B, Grasshoff S, Boemers T, Murphy F, Soylet Y, Dubbers M, Kunst M. Preliminary report on the International Conference for the Development of Standards for the Treatment of Anorectal Malformations. J Pediatr Surg. 2005 Oct;40(10):1521-6. doi: 10.1016/j.jpedsurg.2005.08.002. PMID 16226976
- [Background] Levitt MA, Pena A. Outcomes from the correction of anorectal malformations. Curr Opin Pediatr. 2005 Jun;17(3):394-401. doi: 10.1097/01.mop.0000163665.36798.ac. PMID 15891433
- [Background] Pena A, Devries PA. Posterior sagittal anorectoplasty: important technical considerations and new applications. J Pediatr Surg. 1982 Dec;17(6):796-811. doi: 10.1016/s0022-3468(82)80448-x. PMID 6761417
- [Background] Georgeson KE, Inge TH, Albanese CT. Laparoscopically assisted anorectal pull-through for high imperforate anus--a new technique. J Pediatr Surg. 2000 Jun;35(6):927-30; discussion 930-1. doi: 10.1053/jpsu.2000.6925. PMID 10873037
- [Background] Levitt MA, Kant A, Pena A. The morbidity of constipation in patients with anorectal malformations. J Pediatr Surg. 2010 Jun;45(6):1228-33. doi: 10.1016/j.jpedsurg.2010.02.096. PMID 20620325
- [Background] Levitt MA, Soffer SZ, Pena A. Continent appendicostomy in the bowel management of fecally incontinent children. J Pediatr Surg. 1997 Nov;32(11):1630-3. doi: 10.1016/s0022-3468(97)90470-x. PMID 9396543
- [Background] Rangel SJ, Lawal TA, Bischoff A, Chatoorgoon K, Louden E, Pena A, Levitt MA. The appendix as a conduit for antegrade continence enemas in patients with anorectal malformations: lessons learned from 163 cases treated over 18 years. J Pediatr Surg. 2011 Jun;46(6):1236-42. doi: 10.1016/j.jpedsurg.2011.03.060. PMID 21683229
- [Background] Yong C, Ruo-yi W, Yuan Z, Shu-hui Z, Guang-Rui S. MRI findings in patients with defecatory dysfunction after surgical correction of anorectal malformation. Pediatr Radiol. 2013 Aug;43(8):964-70. doi: 10.1007/s00247-013-2639-8. Epub 2013 Mar 7. PMID 23467755
- [Background] Eltomey MA, Donnelly LF, Emery KH, Levitt MA, Pena A. Postoperative pelvic MRI of anorectal malformations. AJR Am J Roentgenol. 2008 Nov;191(5):1469-76. doi: 10.2214/AJR.07.3773. PMID 18941087
- [Background] Keshtgar AS, Athanasakos E, Clayden GS, Ward HC. Evaluation of outcome of anorectal anomaly in childhood: the role of anorectal manometry and endosonography. Pediatr Surg Int. 2008 Aug;24(8):885-92. doi: 10.1007/s00383-008-2181-1. Epub 2008 May 30. PMID 18512062
- [Background] Caldaro T, Romeo E, De Angelis P, Gambitta RA, Rea F, Torroni F, Foschia F, di Abriola GF, Dall'Oglio L. Three-dimensional endoanal ultrasound and anorectal manometry in children with anorectal malformations: new discoveries. J Pediatr Surg. 2012 May;47(5):956-63. doi: 10.1016/j.jpedsurg.2012.01.051. PMID 22595581
- [Background] Jones MP, Post J, Crowell MD. High-resolution manometry in the evaluation of anorectal disorders: a simultaneous comparison with water-perfused manometry. Am J Gastroenterol. 2007 Apr;102(4):850-5. doi: 10.1111/j.1572-0241.2007.01069.x. PMID 17397410
- [Background] Rintala RJ, Marttinen E, Virkola K, Rasanen M, Baillie C, Lindahl H. Segmental colonic motility in patients with anorectal malformations. J Pediatr Surg. 1997 Mar;32(3):453-6. doi: 10.1016/s0022-3468(97)90604-7. PMID 9094016
- [Background] Zuccarello B, Romeo C, Scalfari G, Impellizzeri P, Montalto AS, D'Oppido D, Campenni A, Formica I, Baldari S. Scintigraphic evaluation of colonic motility in patients with anorectal malformations and constipation. J Pediatr Surg. 2006 Feb;41(2):310-3. doi: 10.1016/j.jpedsurg.2005.11.005. PMID 16481241
- [Background] Demirogullari B, Ozen IO, Karabulut R, Turkyilmaz Z, Sonmez K, Kale N, Basaklar AC. Colonic motility and functional assessment of the patients with anorectal malformations according to Krickenbeck consensus. J Pediatr Surg. 2008 Oct;43(10):1839-43. doi: 10.1016/j.jpedsurg.2008.01.055. PMID 18926217
- [Background] Wexner SD, Marchetti F, Salanga VD, Corredor C, Jagelman DG. Neurophysiologic assessment of the anal sphincters. Dis Colon Rectum. 1991 Jul;34(7):606-12. doi: 10.1007/BF02049902. PMID 2055146
- [Background] Witvliet MJ, Slaar A, Heij HA, van der Steeg AF. Qualitative analysis of studies concerning quality of life in children and adults with anorectal malformations. J Pediatr Surg. 2013 Feb;48(2):372-9. doi: 10.1016/j.jpedsurg.2012.11.018. PMID 23414868
- [Background] Poley MJ, Stolk EA, Tibboel D, Molenaar JC, Busschbach JJ. Short term and long term health related quality of life after congenital anorectal malformations and congenital diaphragmatic hernia. Arch Dis Child. 2004 Sep;89(9):836-41. doi: 10.1136/adc.2002.016543. PMID 15321860
- [Background] Hartman EE, Oort FJ, Visser MR, Sprangers MA, Hanneman MJ, de Langen ZJ, va Heurn LW, Rieu PN, Madern GC, van der Zee DC, Looyard N, van Silfhout-Bezemer M, Aronson DC. Explaining change over time in quality of life of adult patients with anorectal malformations or Hirschsprung's disease. Dis Colon Rectum. 2006 Jan;49(1):96-103. doi: 10.1007/s10350-005-0216-4. PMID 16328611
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Agachan F, Chen T, Pfeifer J, Reissman P, Wexner SD. A constipation scoring system to simplify evaluation and management of constipated patients. Dis Colon Rectum. 1996 Jun;39(6):681-5. doi: 10.1007/BF02056950. PMID 8646957
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Wittrup-Jensen KU, Lauridsen JT, Gudex C et al. Estimating Danish EQ-5D tariffs using TTO and VAS. In: Norinder A, Pedersen K, Roos P, editors. Proceedings of the 18th Plenary Meeting of the EuroQol Group. IHE, The Swedish Institute for Health Economics 2002; 257-292.
- [Background] Obel C, Dalsgaard S, Stax HP, Bilenberg N. [Strengths and Difficulties Questionnaire (SDQ-Dan). A new instrument for psychopathologic screening of children aged 4-16 years]. Ugeskr Laeger. 2003 Jan 27;165(5):462-5. No abstract available. Danish. PMID 12599845
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Donovan JL, Abrams P, Peters TJ, Kay HE, Reynard J, Chapple C, De La Rosette JJ, Kondo A. The ICS-'BPH' Study: the psychometric validity and reliability of the ICSmale questionnaire. Br J Urol. 1996 Apr;77(4):554-62. doi: 10.1046/j.1464-410x.1996.93013.x. PMID 8777617
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Derived] Bjorsum-Meyer T, Christensen P, Baatrup G, Jakobsen MS, Asmussen J, Qvist N. Dyssynergic patterns of defecation in constipated adolescents and young adults with anorectal malformations. Sci Rep. 2020 Nov 12;10(1):19673. doi: 10.1038/s41598-020-76841-5. PMID 33184420
- See also: webpage — http://www.kidscreen.org